CLINICAL TRIAL: NCT07024602
Title: A Phase I, Randomized, Double-blind, Placebo Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Food Effect of ASC50 Tablets in Healthy Adult Participants and Adult Participants With Mild to Moderate Plaque Psoriasis
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Efficacy of ASC50 Tables in Healthy Participants and Participants With Plaque Psoriasis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ascletis Pharma (China) Co., Limited (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASC50-101
Record Dates: First submitted 2025-06-02; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Plaque Psoriasis
Keywords: ASC50; Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- SAD Cohort 1 (Experimental): Participants will receive a single ASC50 (Dose 1) administration or matching placebo
  Interventions: Drug: ASC50 tablets or matching placebo
- SAD Cohort 2 (Experimental): Participants will receive a single ASC50 (Dose 2) administration or matching placebo
  Interventions: Drug: ASC50 tablets or matching placebo
- SAD Cohort 3 (Experimental): Participants will receive a single ASC50 (Dose 3) administration or matching placebo
  Interventions: Drug: ASC50 tablets or matching placebo
- SAD Cohort 4 (Experimental): Participants will receive a single ASC50 (Dose 4) administration or matching placebo
  Interventions: Drug: ASC50 tablets or matching placebo
- SAD Cohort 5 (Experimental): Participants will receive a single ASC50 (Dose 5) administration or matching placebo
  Interventions: Drug: ASC50 tablets or matching placebo
- SAD Cohort 6 (Experimental): Participants will receive a single ASC50 (Dose 6) administration or matching placebo
  Interventions: Drug: ASC50 tablets or matching placebo
- MAD Cohort 1 (Experimental): Participants will receive ASC50 (Dose 1) or matching placebo for 28 days, QD
  Interventions: Drug: ASC50 tablets or matching placebo
- MAD Cohort 2 (Experimental): Participants will receive ASC50 (Dose 2) or matching placebo for 28 days, QD
  Interventions: Drug: ASC50 tablets or matching placebo
- MAD Cohort 3 (Experimental): Participants will receive ASC50 (Dose 3) or matching placebo for 28 days, QD
  Interventions: Drug: ASC50 tablets or matching placebo

INTERVENTIONS:
Drug: ASC50 tablets or matching placebo — Drug: ASC50 administered orally Drug: Placebo administered orally

SUMMARY:
This is a phase I, randomized, double-blind, placebo-controlled, single and multiple ascending dose study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, food effect of ASC50 tablets in healthy adult participants and adult participants with mild to moderate plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants between 18 to 65 years of age inclusive, at the time of screening.
2. Willing and able to give informed consent prior to any study specific procedures being performed.
3. Have venous access sufficient to allow for blood sampling

Exclusion Criteria:

1. Female participants who are pregnant, breastfeeding or plan to be pregnant during the study period and 3 months after last dose.
2. History or presence of any clinically relevant acute or chronic medical or psychiatric condition that could interfere with the subject's safety during the clinical study or expose the subject to undue risk as judged by the Investigator.
3. Have received systemic immunosuppressive therapy (MTX, apremilast, azathioprine, cyclosporine, 6-thioguanine, mercaptopurine, mycophenolate mofetil, hydroxyurea, and tacrolimus) within 4 weeks of first administration of study drug.
4. Have any other conditions, which, in the opinion of the investigator or sponsor, would make the participant unsuitable for inclusion or could interfere with the participant participating in or completing the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Up to Day 7
  Evaluate the incidence of Serious Adverse Events (SAEs) and Adverse Events (AEs)
Adverse Events | Up to Day 43
  Evaluate the incidence of Serious Adverse Events (SAEs) and Adverse Events (AEs)

SECONDARY OUTCOMES:
AUC | Up to Day 7
  Evaluate the Area under the plasma concentration versus time curve of ASC50
AUC | Up to Day 34
  Evaluate the Area under the plasma concentration versus time curve of ASC50
Cmax | Up to Day 7
  Evaluate the Peak Plasma Concentration of ASC50
Cmax | Up to Day 34
  Evaluate the Peak Plasma Concentration of ASC50
T1/2 | Up to Day 7
  Evaluate the Terminal-Phase Half-Life of ASC50
T1/2 | Up to Day 34
  Evaluate the Terminal-Phase Half-Life of ASC50
Tmax | Up to Day 7
  Evaluate the time to reach the maximum concentration of ASC50
Tmax | Up to Day 34
  Evaluate the time to reach the maximum concentration of ASC50
IL-17A | Up to Day 7
  Changes in IL-17A after ASC50 administration
IL-17A | Up to Day 29
  Changes in IL-17A after ASC50 administration
Beta Defensin-2 | Up to Day 29
  Changes in Beta Defensin-2 after ASC50 administration
IL-19 | Up to Day 29
  Changes in IL-19 after ASC50 administration
Psoriasis Area and Severity Index (PASI) | Up to Day 43
  Changes in Psoriasis Area and Severity Index (PASI) after ASC50 treatment.
Target Lesion Severity Score (TLSS) | Up to Day 43
  Changes in Target Lesion Severity Score (TLSS)after ASC50 treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Ascletis Clinical Site, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No